CLINICAL TRIAL: NCT04852991
Title: Modified Purandare's Cervicopexy Versus Abdominal Sacral Hysteropexy as Conservative Surgeries for Genital Prolapse: A Randomized Control Trial
Brief Title: Modified Purandare's Cervicopexy Versus Abdominal Sacral Hysteropexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Elmaraghy, Lecturer of obstetrics and gynecology - faculty of medicine - Ainshams university, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2021-03-28; First posted 2021-04-21 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Purandare cervicopexy (Active Comparator): Apical prolapse will be corrected by Modified Purandare cervicopexy
  Interventions: Procedure: Modified Purandare cervicopexy
- Abdominal sacrohysterpexy (Active Comparator): Apical prolapse will be corrected by Abdominal sacrohysterpexy
  Interventions: Procedure: Abdominal sacral hysteropexy

INTERVENTIONS:
Procedure: Modified Purandare cervicopexy — The modified Purandare's cervicopexy will be performed in low lithotomy position . Pfannenstiel incision was utilized and the abdomen was opened in layers maintaining perfect hemostasis. Uterus will be delivered through the incision and held with uterus holding forceps. The bladder was dissected inferiorly. A 25-30 cm long strip of polypropylene mesh was prepared by soaking. The mesh was fixed anteriorly at the level of isthmus by No.1 polypropylene sutures . The ends of the mesh were brought lateral to rectus muscle retroperitoneally on both sides taking care not to injure the inferior epigastric vessels. After confirming the correct fixation and haemostasis the uterovesical fold of peritoneum was approximated. The ends of the mesh were fixed to the rectus muscle by criss crossing using No. 1 polypropylene sutures. After confirming the haemostasis, the abdomen was closed in layers. Per speculum examination was done to note the reduction of prolapse.
  Arms: Modified Purandare cervicopexy
Procedure: Abdominal sacral hysteropexy — After peritoneal entry through pfannenstiel incision was, the bladder is mobilized off the cervix. Windows are made in the broad ligament at the level of the isthmus. Posteriorly, the rectovaginal space is entered at the level of the uterosacral ligaments. Next, a 15x15-cm polypropylene mesh is used to fashion two 4.5- to 5-cm-wide strips of mesh; one is bisected for a distance of 5 cm to produce a Y-configuration for the anterior mesh.The anterior mesh arms are passed through the broad ligament windows and attached to the cervix and pubocervical fascia using interrupted 2-0 PDS. The posterior mesh is attached to the rectovaginal fascia using transverse-interrupted 2-0 PDS sutures. Once the sacral dissection has exposed the anterior longitudinal ligament, the proximal ends of the 2 mesh strips are attached to the sacral promontory using two 2-0 polyester sutures to provide elevation of the uterus without tension. The peritoneum is closed over the mesh using a 3-0 vicryl suture
  Arms: Abdominal sacrohysterpexy

SUMMARY:
This study aims to compare safety, efficacy and complications of modified Purandare's cervicopexy with abdominal sacral hysteropexy as conservative surgery in the treatment of genital prolapse in reproductive age group patients at Ain Shams Maternity hospital.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP), the herniation of the pelvic organs to or beyond the vaginal walls, is a common condition. Many women with prolapse experience symptoms that impact daily activities, sexual function, and exercise. The presence of POP can have a detrimental impact on body image and sexuality. Nulliparous prolapse is reported to account for 1.5% to 2% of all cases of genital prolapse . The incidence rises to 5 -8 % for young women who have delivered one or two children. As this type of prolapse occurs at a younger age, the surgical technique should not only reduce the prolapse but also retain the reproductive function. Various conservative surgeries have been described in the past, each having their own merits and de-merits .

Pelvic organ prolapse (POP) is affecting women of all ages. Epidemiological studies suggest a lifetime risk of prolapse or incontinence surgery of between 7 and 19% . In an ageing population, the incidence of these surgeries would only be expected to increase, although the increasing Caesarean Section rates and smaller family size in recent years will have a negative impact on the prevalence of these conditions. There are many approaches to the surgical correction of POP, which frequently reflect the nature and anatomical site of the defective support, but essentially the surgeon has to decide whether to perform this surgery vaginally or via the abdomen as an open or laparoscopic procedure. If performed vaginally, further decisions regarding the use of synthetic or biological graft to reinforce the repair need to be made.

The core of the modified purandare's cervicopexy is fixation of the uterine isthmus by a 25-30 cm long strip of polypropylene mesh to the rectus muscle by criss crossing using No. 1 polypropylene sutures.

Modified purandare's cervicopexy is easy to perform and provides dynamic support to the uterus, improves fertility, doesn't interfere with vaginal birth and if caesarean delivery is required doesn't damage the mesh thus reducing the recurrence of prolapse and has many advantages compared to the original operation which can favourably affect the outcome, such as: criss crossing of mesh on rectus muscle which provides a space for low transverse incision for caesarean section without compromising the mesh anchoring and retaining the support. This surgery is technically easy to perform and complications like Periosteitis, ureteric and sigmoid injuries are avoided.

Abdominal sacral hysteropexy remains a viable alternative for women undergoing pelvic reconstructive surgery who wish to retain their uteri, providing comparable rates of overall improvement and symptom change. Avoiding hysterectomy decreases the risk of mesh erosion but may increase the risk of subsequent recurrent prolapse, specifically in the anterior compartment.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 20 years - 40 years
2. BMI: 20 to 35 kg\m2
3. Any parity with desire for future pregnancy

Exclusion Criteria:

1. 1st degree uterine prolapse.
2. Previous correction of apical prolapse.
3. Co-existing uterine pathology e.g. uterine fibroid .

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Recurrence | twelve months after the procedure
  After the procedure there will be follow up visits at 12 months respectively to detect if there is recurrence or not by history taking and pelvic examination.

SECONDARY OUTCOMES:
Operative time | In minutes from skin incision till closure of the skin and excluding time of concomitant surgical procedures.
  Total operative time from skin incision till closure of the skin and excluding time of concomitant surgical procedures.
Intra operative blood loss | During the procedure
  Intraoperative blood loss will be estimated via:
  * Amount of blood in suction bottle.
  * Estimation based on the number of soaked gauzes by weighing the gauzes used in the procedure before and after surgery ( each 1 mg f corresponds to 1 ml of blood)
  * Drop in postoperative hemoglobin and hematocrit when compared with preoperative values
Need for blood transfusion | During the procedure
  number of participants who need blood transfusion
Postoperative pain the linear 10cm visual analogue scale. Range is from 10(unbearable pain) to zero (no pain) | This will be assessed after 6 hours, 12 hours and 24 hours from the operation
  - Postoperative pain will be assessed using the linear 10cm visual analogue scale. Range is from 10(unbearable pain) to zero (no pain).
Duration of post operative hospital stay. | immediately surgery
  Duration of postoperative hospital stay will be measured from the end of the procedure till discharge from hospital and it will be measured in hours
Bowel injury | During the procedure
  number of participants who suffered from bowel injury during the procedure
Vascular injury | During the procedure
  number of participants who suffered from vascular injury during the procedure
Subfascial hematoma | up to 6 weeks after surgery
  number of participants who will suffer from subfascial hematoma
urinary tract infection | up to 6 weeks after surgery
  number of participants who will suffer from urinary tract infection
Surgical site infection | up to 6 weeks after surgery
  number of participants who will suffer from surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Nasr Eldeen, MD, Study Director — AinShams university
Locations (1):
- AinShams university maternity hospital, Cairo, Egypt

REFERENCES:
- [Background] Lowder JL, Ghetti C, Nikolajski C, Oliphant SS, Zyczynski HM. Body image perceptions in women with pelvic organ prolapse: a qualitative study. Am J Obstet Gynecol. 2011 May;204(5):441.e1-5. doi: 10.1016/j.ajog.2010.12.024. Epub 2011 Feb 2. PMID 21292234
- [Background] Virkud A. Conservative Operations in Genital Prolapse. J Obstet Gynaecol India. 2016 Jun;66(3):144-8. doi: 10.1007/s13224-016-0909-8. Epub 2016 Apr 29. PMID 27298521
- [Background] R., Rameshkumar & Kamat, Leena & Tungal, Spoorthi & Moni, Suma. (2017). Modified purandare's cervicopexy-a conservative surgery for genital prolapse: a retrospective study. International Journal of Reproduction, Contraception, Obstetrics and Gynecology. 6. 10.18203/2320-1770.ijrcog20171529.
- [Background] Smith FJ, Holman CD, Moorin RE, Tsokos N. Lifetime risk of undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 2010 Nov;116(5):1096-100. doi: 10.1097/AOG.0b013e3181f73729. PMID 20966694
- [Background] Cvach K, Dwyer P. Surgical management of pelvic organ prolapse: abdominal and vaginal approaches. World J Urol. 2012 Aug;30(4):471-7. doi: 10.1007/s00345-011-0776-y. Epub 2011 Oct 22. PMID 22020436
- [Background] Cvach K, Geoffrion R, Cundiff GW. Abdominal sacral hysteropexy: a pilot study comparing sacral hysteropexy to sacral colpopexy with hysterectomy. Female Pelvic Med Reconstr Surg. 2012 Sep-Oct;18(5):286-90. doi: 10.1097/SPV.0b013e3182673772. PMID 22983272
- [Background] • Cvach, K. and Cundiff, G. Abdominal Sacral Hysteropexy: Clinical Outcomes Compared to Abdominal Sacral Colpopexy With Concurrent Hysterectomy. Univers. British Columbia (UBC), 2008, 677-678.
- [Background] Lapaire O, Schneider MC, Stotz M, Surbek DV, Holzgreve W, Hoesli IM. Oral misoprostol vs. intravenous oxytocin in reducing blood loss after emergency cesarean delivery. Int J Gynaecol Obstet. 2006 Oct;95(1):2-7. doi: 10.1016/j.ijgo.2006.05.031. Epub 2006 Aug 23. PMID 16934269
- [Background] Hawksley H. Pain assessment using a visual analogue scale. Prof Nurse. 2000 Jun;15(9):593-7. PMID 11129939